CLINICAL TRIAL: NCT03734939
Title: Health and Cardiovascular Risk Factors Survey in the 31's Slum.
Brief Title: Health and Cardiovascular Risk Factors in Slums.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacion GESICA (Other)
Collaborators: Escuela de Psicología Social Pichon Riviere (Unknown); Corriente Salvador Maza (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0004
Record Dates: First submitted 2018-10-11; First posted 2018-11-08 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases
Keywords: cardiovascular risk factor; Slums; survey; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None intervention is planned. — None intervention is planned, just a survey.

SUMMARY:
Cardiovascular risk factors and disease burden has been showed to affect more deeply to poorer populations. People who live in slums are the most vulnerable subgroup in the populations where, paradoxically scarcity of data exists on risk factors and cardiovascular disease burden.

Our study aim to describe the prevalence of cardiovascular risk factors and cardiovascular disease burden in a representative sample of an urban slum of Buenos Aires city, using validated questions from the National Risk Factors Survey (edition 2013). Also, the investigators will measure blood pressure and cardiac rate to all study participants.

DETAILED DESCRIPTION:
Cardiovascular risk factors and disease burden has been showed to affect more deeply to poorer populations. People who live in slums are the most vulnerable subgroup in the populations where, paradoxically scarcity of data exists on risk factors and cardiovascular disease burden.

Hypothesis: the prevalence of modifiable cardiovascular risk factors in an urban slum from Buenos Aires city is higher than the rest of the country and, consequently requires a distinctive management approach.

Objectives:

1. To measure the prevalence of cardiovascular risk factors in a representative sample of the villa 31 (an urban slum from Buenos Aires city).
2. To measure the self-perceived health in a representative sample of the villa 31 (urban slum from Buenos Aires city).

Design: observational study. Survey. Procedures: the survey will be conducted by neighbors from the slum that received specific training as community health workers and were trained on the use of the survey questionnaire and for blood pressure measuring.

Sampling: representative samples of slum population will be obtained using probabilistic, multi-staged sampling methods.

Blood pressure measures: blood pressure will be measured using automatic blood pressure monitoring device with appropriate cuff sizes.

Statistical analyses: categorical variables will be expressed as numbers and percentages, and continuous variable as means and standard deviations or medians and interquartile ranges. Between groups comparisons will be conducted using chi2 test for categorical variables and T test or Mann-Whitney U's test for continuous variables. To compare the prevalence of risk factors with the rest of the country, the database will be jointed with the national risk factor survey (publicly available). All analyses will be weighted to account for the sampling method.

ELIGIBILITY:
Inclusion Criteria: >= 18 years. Sign the informed consent.

-

Exclusion Criteria: Unable to answer the survey. Unwilling to participate.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults of the slum that accept to participate in the survey.
Sampling Method: Probability Sample
Enrollment: 2265 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Hypertension | Through study completion, an average of 3 months
  Blood pressure >=140/90 mmHg or being taking antihypertensive medication.
Smoking | Through study completion, an average of 3 months
  Percentage of participants that self-report current smoking
Hypercholesterolemia | Through study completion, an average of 3 months
  Self-reported plasma high cholesterol levels.
Diabetes | Through study completion, an average of 3 months
  Percentage of participants that self-report as had been diagnosed as diabetic or receiving medical therapy for diabetes.
Self-perceived health | Through study completion, an average of 3 months
  Percentage of participants that report their health status as self-perceived in a 5-points Likert' scale from "Excellent" to "Bad"

SECONDARY OUTCOMES:
Previous myocardial infarction | through study completion, an average of 3 months
  Self-reported history of myocardial infarction.
Previous stroke | through study completion, an average of 3 months
  Self-reported history of stroke.
Physical activity | Through study completion, an average of 3 months
  Percentage of participants with self-reported physical activity levels in a Likert' scale (from "Less than 10 min/week" to "Equal or more than 150 min/week").
Healthy diet | through study completion, an average of 3 months
  Self-reported consumption of vegetables and fruits.
Body mass index | through study completion, an average of 3 months
  Body weight divided by the height squared in meters (both body weight and height as self-reported.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Mariani, MD, Principal Investigator — Fundación GESICA
Locations (1):
- Fundación GESICA, Ciudad Autónoma de Buenos Aire, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No